CLINICAL TRIAL: NCT04878484
Title: A Phase 1 Open-label Study to Evaluate the Safety, Tolerability, and Activity of TCRT-ESO-A2 Autologous T Cells Expressing TCR Specific for NY-ESO-1 in Subjects With Advanced Solid Tumors
Brief Title: Evaluate TCRT-ESO-A2 Autologous T Cells Expressing TCR Specific for NY-ESO-1 in Subjects With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AX TCRT 001
Record Dates: First submitted 2021-03-01; First posted 2021-05-07 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumor
Keywords: NY-ESO-1

STUDY DESIGN:
Intervention Model Description: open-label, multi-site, "3+3" dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: TCRT-ESO-A2: 0.3 × 1010 TCRT-ESO-A2 cells * ±30% (Experimental): Subjects will be evaluated for DLTs up to 28 days post-TCRT-ESO-A2 infusion. Enrollment into a dose level will be suspended if two of no more than six subjects at a dose level experience dose-limiting toxicity. Prior to increasing the dose, a cohort management meeting will be held after the final enrolled subject has been followed for up to28 days. The decision to increase to the next dose level will be a joint decision of the clinical site Investigators and Sponsor. At each cohort, there will be at least 7 days between infusion of each subject in the cohort.
  Interventions: Biological: TCRT-ESO-A2
- Cohort 2: TCRT-ESO-A2: 1.0 × 1010 TCRT-ESO-A2 cells ±30% (Experimental): Subjects will be evaluated for DLTs up to 28 days post-TCRT-ESO-A2 infusion. Enrollment into a dose level will be suspended if two of no more than six subjects at a dose level experience dose-limiting toxicity. Prior to increasing the dose, a cohort management meeting will be held after the final enrolled subject has been followed for up to28 days. The decision to increase to the next dose level will be a joint decision of the clinical site Investigators and Sponsor. At each cohort, there will be at least 7 days between infusion of each subject in the cohort. The decision to increase to the next dose level will be a joint decision of the clinical site Investigators and Sponsor.
  Interventions: Biological: TCRT-ESO-A2
- Cohort 3: TCRT-ESO-A2 : 3.0 × 1010 TCRT-ESO-A2 cells ±30% (Experimental): Subjects will be evaluated for DLTs up to 28 days post-TCRT-ESO-A2 infusion. Enrollment into a dose level will be suspended if two of no more than six subjects at a dose level experience dose-limiting toxicity. Prior to increasing the dose, a cohort management meeting will be held after the final enrolled subject has been followed for up to28 days. The decision to increase to the next dose level will be a joint decision of the clinical site Investigators and Sponsor. At each cohort, there will be at least 7 days between infusion of each subject in the cohort.
  Interventions: Biological: TCRT-ESO-A2

INTERVENTIONS:
Biological: TCRT-ESO-A2 — TCRT-ESO-A2 is an autologous cell therapy comprised of a subject's T cells stimulated ex vivo and transduced with a lentiviral vector encoding an affinity enhanced TCR targeting tumor-associated antigen NY-ESO-1.

SUMMARY:
TCRT-ESO-A2 is an autologous cell therapy comprised of a subject's T cells stimulated ex vivo and transduced with a lentiviral vector encoding an affinity enhanced TCR targeting tumor-associated antigen NY-ESO-1.

This study will investigate the safety, tolerability, activity, and pharmacokinetics/ pharmacodynamics of TCRT-ESO-A2 infusion. A maximum tolerated dose study of TCRT-ESO-A2 in subjects with advanced malignancies expressing NY-ESO-1 is considered to be an acceptable risk. Once safety, tolerability, and pharmacokinetic/pharmacodynamic data are available, the activity of TCRT-ESO-A2 in NY-ESO-1-positive tumors may be explored further.

DETAILED DESCRIPTION:
This is a Phase 1 open-label, multi-site, "3+3" dose escalation, study to evaluate the maximum tolerated dose, safety and tolerability, of TCRT-ESO-A2 suspension for IV infusion. Approximately 24 HLA-A*0201-positive subjects with head and neck cancer, hepatocellular carcinoma, lung squamous cell carcinoma, synovial sarcoma, and triple-negative breast cancer expressing NY-ESO-1 who have received at least first-line therapy for their cancer, or which there is no accepted therapy will be enrolled. Tumor tissue samples will be evaluated and scored using the NY-ESO-1 IHC assay developed specifically to support this study.

Following screening and enrollment (approximately Days -63 to -36) subjects will undergo leukapheresis for T cell collection at approximately Day -35 (Figure 3). Harvested cells will be fractionated, genetically engineered, and expanded ex vivo to produce autologous TCRT-ESO-A2 TCR-T. Following TCRT-ESO-A2 product release, subjects will receive a 3-day, non-myeloablative lymphodepletion regimen of fludarabine/cyclophosphamide from approximately Days -5 to -3 (recommend Wednesday to Friday) to prime the subject for immune re-population. Subjects will receive their TCRT-ESO-A2 cell product on Day 1 (recommend Monday) as an IV infusion over approximately 30 minutes. Within 30 minutes after completion of TCRT-ESO-A2 infusion, low dose subcutaneous aldesleukin (rhIL-2) will be administered at 500,000 IU BID daily for 14 days.

Dose escalation will be divided into three dose groups of three subjects each, with doses calculated as the number of TCR Vβ8-positive cells (total TCRT-ESO-A2 dose), with an allowable variance in cell count of ±30%. Escalation to higher doses will be based on the safety and tolerability of the previous cohort evaluated. If dose-limiting toxicity is observed in one subject at a dose level, up to an additional three dose limiting toxicity-evaluable subjects will be enrolled at that dose level. Subjects will be evaluated for dose limiting toxicity up to 28 days post-TCRT-ESO-A2 infusion. Prior to increasing the dose, a cohort management meeting will be held after the final enrolled subject has been followed for up to 28 days. The decision to increase to the next dose level will be a joint decision of the clinical site Investigators and Sponsor. At each cohort, there will be at least 7 days between infusion of each subject in the cohort. Enrollment into a dose level will be suspended if two of no more than six subjects at a dose level experience dose-limiting toxicity.

Three dose groups of subjects will be enrolled:

Cohort 1: 0.3 × 1010 TCRT-ESO-A2 cells* Cohort 2: 1.0 × 1010 TCRT-ESO-A2 cells* Cohort 3: 3.0 × 1010 TCRT-ESO-A2 cells*

* ±30% Subjects will be monitored daily during in-patient hospitalization for 5 days post dose. Subjects will then visit an out-patient clinic weekly during the Dose Limiting Toxicity Evaluation Period of 4 weeks and followed at approximately Days 60, 90, and every 3 months until confirmation of disease progression. Disease monitoring will be conducted by Magnetic Resonance Imaging or Computed Tomography scan (as appropriate for disease), during screening (if recent scans are not available), during lead-in approximately 7 days prior to TCRT-ESO-A2 infusion, at approximately Days 28, 60, 90, and every 3 months until confirmation of disease progression. If subjects remain clinically stable, confirmation of progression may be assessed 4- to 8-weeks later. Positron emission tomography scanning may be used as appropriate as an adjunct. Tumor biopsies will be taken from non-target lesions, if accessible, at baseline, approximately Days 28, 90, 180, and upon progression. Ascites/pleural fluid may be collected in addition to biopsies for correlative research studies if the subject requires paracentesis or pleuracentesis. At progression, long term follow-up will commence. During long term follow-up, subjects will be followed twice yearly for up to 5 years post-infusion and then annually for up to 15 years.

Timing of tumor and liquid biopsies may be adjusted as may the timing of other procedures or safety studies. In addition, up to 150 additional mL of blood may be collected over a three-month period without amendment of the protocol. Additional safety measures may be included, and tests may be done at any time if clinically indicated. In addition, if objective responses are observed in tumors after the safety of each cohort has been evaluated, up to 12 additional subjects with that tumor type (up to 2 tumor types) may be enrolled to further explore the tumor response rate in that tumor type.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign an informed consent form (ICF).
2. Age ≥18 years of age at the time of informed consent.
3. HLA-A*0201 positive by high resolution testing.
4. Any of the following solid tumors with positive NY-ESO-1 expression characterized by IHC:

   1. Head and neck cancer with ≥85% of tumor cells scored ≥1+.
   2. Hepatocellular carcinoma with ≥20% of tumor cells scored ≥1+.
   3. Lung squamous cell carcinoma with ≥20% of tumor cells scored ≥1+.
   4. Synovial sarcoma with ≥65% of cells scored ≥1+.
   5. Triple-negative breast cancer with ≥20% of cells scored ≥1+.
5. Received standard curative or palliative therapy including any targeted therapy based on mutation status for their cancer, or advanced solid tumors for which there is no accepted therapy, standard therapies are no longer effective, or the subject refuses additional standard therapy.
6. Measurable disease as defined per RECIST 1.1 (Eisenhauer 2009).
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
8. Life expectancy of >4 months.
9. Adequate hematologic status as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) to maintain:

   1. White blood cell count ≥3,000/mcL.
   2. Absolute neutrophil count ≥1,000/mcL.
   3. Platelet count ≥100,000/mcL.
   4. Hemoglobin ≥9.0 g/dL.
10. Adequate liver function as demonstrated by:

    1. Serum alanine transaminase (ALT) and aspartate transaminase (AST) ≤3 × upper limit of normal, except in subjects with liver metastasis, who must have AST and ALT ≤5 × upper limit of normal.
    2. Total bilirubin ≤1.5 × upper limit of normal, except in subjects with Gilbert's Syndrome, who must have total bilirubin ≤3.0 × upper limit of normal.
11. Creatinine clearance ≥50 mL/min. Creatinine clearance of subjects <65 years of age may be estimated by the Cockcroft-Gault formula. Subjects ≥65 years of age must have renal function measured either by 24-hour urine creatinine collection or by nuclear medicine glomerular filtration rate.
12. Prior therapies:

    1. Targeted or immunotherapy must be completed at least 4 weeks prior to leukapheresis.
    2. Chemotherapy must be completed at least 3 weeks prior to leukapheresis.
    3. Systemic corticosteroid or other immunosuppressive therapy must be completed at least 2 weeks prior to leukapheresis.
13. Recovered from previous surgery or treatment-related adverse reactions to <grade 2 CTCAE (except for toxicities such as alopecia or vitiligo or toxicities that may be permanent such as neuropathy) prior to lymphodepletion chemotherapy.
14. Men who are sterile (including vasectomy confirmed by post vasectomy semen analysis) or agree to use a condom with spermicide and to not donate sperm during the study and until the persistence of TCRT-ESO-A2 is no longer detected by qPCR or up to 15 years.
15. Women of non-child bearing potential due to surgical sterilization (at least 6 weeks following surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history or menopause (i.e., no menstrual bleeding for more than 12 months in a woman aged ≥45 years), OR women of childbearing potential who test negative for pregnancy at Screening based on serum pregnancy test must be using a highly effective method of contraception from the time of Screening until the persistence of TCRT-ESO-A2 is no longer detected by qPCR or up to 15 years. Note: Highly effective methods of contraception that result in a low failure rate (i.e., <1% per year) when used consistently and correctly include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or sexual abstinence. True abstinence, when in line with the preferred and usual lifestyle of the subject, is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of study participation and until the persistence of TCRT-ESO-A2 is no longer detected by qPCR. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, and post-ovulation method) and withdrawal are not acceptable methods of contraception.

5.3 Exclusion Criteria

Eligible subjects must not have/be:

1. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease or AIDS).
2. Known allergic reactions to any component of the treatments in this study.
3. Echocardiography (ECHO) or multigated acquisition scan (MUGA) indicative of left ventricular ejection fraction (LVEF) ≤45%.

Exclusion Criteria:

* Eligible subjects must not have/be:

  1. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease or AIDS).
  2. Known allergic reactions to any component of the treatments in this study.
  3. Echocardiography (ECHO) or multigated acquisition scan (MUGA) indicative of left ventricular ejection fraction (LVEF) ≤45%.
  4. Pulmonary function test of forced expiratory volume in the first second (FEV1) ≤60% in subjects with a prolonged history of cigarette smoking (e.g. ≥20 pack-year smoking history).
  5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements.
  6. Subjects with infection requiring treatment, including but not limited to active tuberculosis, COVID-19, known HIV positive subjects or subjects with clinically active hepatitis A, B and C.
  7. Planning to take the following medications within 4 weeks of TCRT-ESO-A2 infusion or during the study: long-term systemic use of steroid hormones, hydroxyurea, immunomodulatory drugs (such as interleukin 2, interferon α or γ, GM-CSF, mTOR inhibitor, cystatin, thymosin, etc.). Recent use of inhaled or topical steroids, topical 5-fluorouracil is not exclusionary, however, use of inhaled steroids before leukapheresis and blood draws should be discouraged.
  8. Untreated or symptomatic brain metastasis.
  9. History of organ transplantation or allogeneic stem cell transplantation.
  10. Known uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease or liver failure.
  11. Previous use of any gene therapy product.
  12. Not suitable for enrollment at the discretion of the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Evaluate up to Eighteen Subjects With Tumors Expressing TCRT-ESO-A1 and Having Dose Limiting Toxicity Adverse Events as Assessed by CTCAE-Version 5 | Day 28
  TCRT-ESO-A2 maximum tolerated dose as assessed by the occurrence of dose-limiting toxicity adverse events at least possibility related to TCRT-ESO - A2 in two of six subjects who received TCRT-ESO-A2

SECONDARY OUTCOMES:
Dose Escalation: Tumor Response for Partial Response as Assessed by RECIST 1.1. | Day 28 and every 3 months until disease progression averaging one year
  Evaluate tumor response for partial response response as assessed by RECIST 1.1, standardized assessment with complete response being the highest and disease progression being the lowest outcome.
Dose Escalation: Tumor Response Stable Disease as Assessed by RECIST 1.1. | Day 28 and every 3 months until disease progression averaging one year
  Evaluate tumor response for stable disease response response as assessed by RECIST 1.1, a standardized assessment with complete response being the highest and disease progression being the lowest outcome.
Dose Escalation: Tumor Response Disease Progression as Assessed by RECIST 1.1. | Day 28 and every 3 months until disease progression averaging one year
  Evaluate tumor response for disease progression response as assessed by RECIST 1.1, a standardized assessment with complete response being the highest and disease progression being the lowest outcome.
Dose Escalation: Tumor Response Overall Survival as Assessed by RECIST 1.1. | Day 28 and every 3 months until disease progression averaging one year
  Evaluate tumor response for overall survival as assessed by RECIST 1.1, a standardized assessment with complete response being the highest and disease progression being the lowest outcome.
Dose Escalation: Tumor Response Progression-Free Survival as Assessed by RECIST 1.1. | Day 28 and every 3 months until disease progression averaging one year
  Evaluate tumor response for disease progression-free survival as assessed by RECIST 1.1, a standardized assessment with complete response being the highest and disease progression being the lowest outcome.
Dose Escalation: Persistence of Genetically Modified T Cells in Vivo and T Cell Subpopulations | Day 28 to disease progression averaging one year
  Evaluate the persistence of genetically modified T cells in vivo as assessed by evidence of an abundance of T cell subpopulations in circulation
Dose Escalation: Persistence of Genetically Modified T Cells in Vivo and Antigen Specific CD8 + Cytotoxic T lymphocytes | Day 28 to disease progression averaging one year
  Evaluate persistence of genetically modified T cells in vivo and antigen specific CD8 + cytotoxic T lymphocytes in circulation
Dose Escalation: Phenotype of Genetically Modified T Cells in Vivo and Functional Characteristics | Day 28 to disease progression averaging one year
  Evaluate the phenotype of genetically modified T cells in vivo as assessed by functional characteristics
Dose Escalation: Monitor Presence of Potentially Replication-Competent Lentivirus before TCRT ESO A2 Infusion | Days - 7
  Monitor presence of potentially Replication-Competent Lentivirus before TCRT 001 ESO A2 infusion as assessed by qualitative PCR assay to detect and measure gene coding copies for the VSV- G Envelope Protein
Dose Escalation: Monitor Presence of Potentially Replication-Competent Lentivirus After TCRT ESO A2 Infusion | Days 90 and 270
  Monitor presence of potentially Replication-Competent Lentivirus after TCRT 001 ESO A2 infusion as assessed by qualitative PCR assay to detect and measure gene coding copies for the VSV- G Envelope Protein
Maximum Tolerated Dose Expansion: Overall Survival Assessment | Baseline to disease progression averaging one year
  Evaluate overall survival as assessed by RECIST 1.1
Maximum Tolerated Dose Expansion: Objective Response Rate Assessment | 3 months
  Evaluate objective response rate as assessed by RECIST 1.1
Maximum Tolerated Dose Expansion: Progression-free Survival Assessment | 3 months
  Evaluate progression-free survival 3-months as assessed by RECIST 1.1 every 3 months
Maximum Tolerated Dose Expansion: Disease Control Rate Assessment | 3 months
  Evaluate disease control rate at 3-months as assessed by RECIST 1.1
Maximum Tolerated Dose Expansion: TCRT-ESO-A2 Maximum Concentration Pharmacokinetic Characteristics | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year
  Evaluate TCRT-ESO-A2 as assessed by CD3-Positive/Tetramer-Positive T Cells maximum concentration
Maximum Tolerated Dose Expansion: TCRT-ESO-A2 Maximum Concentration pharmacokinetic characteristics | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year
  Evaluate TCRT-ESO-A2 as assessed by CD3-Positive/Tetramer-Positive T Cells Time to maximum concentration
Maximum Tolerated Dose Expansion: TCRT-ESO-A2 Half-Life pharmacokinetic characteristic | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year
  Evaluate TCRT-ESO-A2 as assessed by CD3-positive/tetramer-positive T Cells Half-Life
Maximum Tolerated Dose Expansion: TCRT-ESO-A2 time last pharmacokinetic characteristic | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year
  Evaluate TCRT-ESO-A2 as assessed by CD3-positive/tetramer-positive T Cells
Maximum Tolerated Dose Expansion: Evaluate Tumor for Complete Response as Assessed by RECIST 1.1. | Baseline to disease progression averaging one year
  Evaluate tumor for complete response as assessed by RECIST 1.1, a standardized assessment with complete response the highest and disease progression the lowest outcome assessment
Maximum Tolerated Dose Expansion: Evaluate Tumor for Partial Response as Assessed by RECIST 1.1. | Baseline to disease progression averaging one year
  Evaluate tumor for partial response as assessed by RECIST 1.1, a standardized assessment with complete response the highest and disease progression the lowest outcome assessment
Maximum Tolerated Dose Expansion: Evaluate Tumor for Stable Disease as Assessed by RECIST 1.1. | Baseline to disease progression averaging one year
  Evaluate tumor for stable disease response as assessed by RECIST 1.1, a standardized assessment with complete response the highest and disease progression the lowest outcome assessment
Maximum Tolerated Dose Expansion: Evaluate Tumor for Disease Progression as Assessed by RECIST 1.1. | Baseline to disease progression averaging one year
  Evaluate tumor for disease progression as assessed by RECIST 1.1, a standardized assessment with complete response the highest and disease progression the lowest outcome assessment
Maximum Tolerated Dose Expansion: Evaluate Tumor for Progression-Free Survival as Assessed by RECIST 1.1. | Baseline to disease progression averaging one year
  Evaluate tumor for progression-free survival as assessed by RECIST 1.1, a standardized assessment with complete response the highest and disease progression the lowest outcome assessment
Maximum Tolerated Dose Expansion: Evaluate Tumor for Overall Survival as Assessed by RECIST 1.1. | Baseline to disease progression averaging one year
  Evaluate tumor for overall survival as assessed by RECIST 1.1, a standardized assessment with complete response the highest and disease progression the lowest outcome assessment
Maximum Tolerated Dose Expansion: Persistence of Genetically Modified T Cells in Vivo as Assessed by Functional Characteristics and Persistence in the Circulation | Baseline to disease progression averaging one year
  Evidence of abundance of T cell subpopulations, antigen specific CD8+ cytotoxic T lymphocytes , functional characteristics and persistence in the circulation
Maximum Tolerated Dose Expansion: Monitor Presence of Potentially Replication-Competent Lentivirus (RCL) before TCRT ESO A2 Infusion | Day -7
  Monitor presence of potentially Replication-Competent Lentivirus before TCRT 001 ESO A2 infusion as assessed by qualitative PCR assay to detect and measure gene coding copies for the VSV- G Envelope Protein
Maximum Tolerated Dose Expansion: Monitor Presence of Potentially Replication-Competent Lentivirus (RCL) after TCRT ESO A2 Infusion | Days 90, 270
  Monitor presence of potentially Replication-Competent Lentivirus after TCRT 001 ESO A2 infusion as assessed by qualitative PCR assay to detect and measure gene coding copies for the VSV- G Envelope Protein
Long Term Follow Up Period: Monitor VSV-G DNA qualitative PCR | Progression of disease up to 15 years
  Monitor presence of potentially Replication-Competent Lentivirus as assessed by qualitative PCR assay to detect and measure gene coding copies for the VSV- G Envelope Protein
Long Term Follow Up Period: Monitor New Incidence of Potentially Product-Related Infection | Progression of disease up to 15 years
  Monitor new incidence of potentially product-related infection as assessed by annual or biannual long term follow-up interview
Long Term Follow Up Period: Monitor New Incidence of malignancy | Progression of disease up to 15 years
  Monitor incidence of new malignancy(ies) as reported in annual or biannual long term follow-up interview

OTHER OUTCOMES:
Explore Persistence of Genetically Modified T cells in vivo. | Baseline to disease progression averaging one year
  Characteristics of Persistence of Genetically Modified T cells in vivo will be assessed by multiple linear regression.
Explore Phenotype of Genetically Modified T cells in vivo. | Baseline to disease progression averaging one year
  Characteristics of phenotype of genetically modified T cells in vivo will be assessed by multiple linear regression.
Explore Presence of CA-125 Tumor Immune Biomarker Before TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of CA-125 tumor biomarker before TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Presence of CA-125 Tumor Immune Biomarker after TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of CA-125 Tumor Biomarker After TCRT-ESO-A2 Infusion will be assessed by multiple linear regression.
Explore Presence of CEA Tumor Immune Biomarker Before TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of CEA tumor immune biomarker before TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Presence of CEA Tumor Immune Biomarker After TCRT-ESO-A2 infusion | Baseline to disease progression averaging one year
  The presence of CEA tumor immune biomarker after TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Presence of PSA Tumor Immune Biomarker Before TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of PSA tumor biomarker before TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Presence of PSA Tumor Immune Biomarker After TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of PSA tumor biomarker after TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Distribution of PSA Tumor immune Biomarker After TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The distribution of PSA tumor biomarker after TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Cytokine IFN-γ Presence Before TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of systemic cytokine IFN-γ before TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Cytokine IFN-γ Presence After TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of systemic cytokine IFN-γ after TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Presence of Targeted Antigen NY-ESO-1, Before TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  The presence of targeted antigen NY-ESO-1 before TCRT-ESO-A2 infusion Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months will be assessed by multiple linear regression.
Explore Presence of Targeted Antigen NY-ESO-1 After TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  Evaluate the presence and distribution of and targeted antigen NY-ESO-1 after TCRT-ESO-A2 infusion
Explore Distribution of Targeted Antigen NY-ESO-1 After TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  Evaluate the distribution of targeted antigen NY-ESO-1 after before TCRT-ESO-A2 infusion will be assessed by multiple linear regression.
Explore Presence of PSA Tumor Immune Biomarker | Baseline to disease progression averaging one year
  The presence of PSA tumor biomarker will be assessed by multiple linear regression.
Explore Presence of CEA Tumor Immune Biomarker | Baseline to disease progression averaging one year
  The presence of CEA tumor biomarker will be assessed by multiple linear regression.
:Explore Persistence of Genetically Modified T cells in vivo. | Baseline to disease progression averaging one year
  Characteristics of persistence of genetically modified T cells in vivo will be assessed by multiple linear regression.
Explore Evaluate Presence of Cytokine IFN-γ MTD Expansion: Evaluate cytokine IFN-γ before and after TCRT-ESO-A2 infusion | Baseline to disease progression averaging one year
  The presence of systemic cytokine IFN-y will be assessed by multiple linear regression
Explore Evaluate Cytokine IFN-γ Before TCRT-ESO-A2 Infusion MTD Expansion: Evaluate cytokine IFN-γ before and after TCRT-ESO-A2 infusion | Baseline to disease progression averaging one year
  Evaluate the presence of systemic cytokine IFN-y before TCRT-ESO-A2 infusion will be assessed by multiple linear regression
Explore Presence of Targeted Antigen NY-ESO-1 Before TCRT-ESO-A2 Infusion | Baseline to disease progression averaging one year
  Evaluate the presence of targeted antigen NY-ESO-1, before TCRT-ESO-A2 infusion will be assessed by multiple linear regression
Explore Perform NY-ESO-1 Immunohistochemistry Assay Using a Four-point Semi-quantitative Scale (low to high): 0, 1+, 2+, 3+ With High Inferring a Better Outcome | Baseline to disease progression averaging one year
  Evaluate the subject tumor to determine cut-off high and low NY ESO - 1 expression.
Explore Association Between Maximum TCRT ESO A2 Concentration time and Systemic Cytokine IFN-γ Level | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year.
  The association between maximum TCRT ESO A2 concentration time and systemic cytokine IFN-γ level will be assessed by multiple linear regression.
Explore Association Between Maximum TCRT ESO A2 Concentration time and Systemic Cytokine IL-6 Level | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year.
  The association between maximum TCRT ESO A2 concentration time and systemic cytokine IL-6 level will be assessed by multiple linear regression.
Explore Association Between Maximum TCRT ESO A2 Concentration time and Systemic Cytokine TNFα Level | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year.
  The association between maximum TCRT ESO A2 concentration time and systemic cytokine IFN-γ level will be assessed by multiple linear regression.
Explore Association Between Maximum Dose Concentration Time and Disease Appropriate Circulating Tumor Marker CA-125 | Day 28
  The association between pharmacokinetic maximum dose concentration time and pharmacodynamic disease appropriate circulating tumor marker CA-125 will be assessed by multiple linear regression.
Explore Association Between Pharmacokinetic Maximum Dose Concentration Time and Disease Appropriate Circulating Tumor Marker CEA | Day 28
  The association between pharmacokinetic maximum dose concentration time and pharmacodynamic disease appropriate circulating tumor marker CEA will be assessed by multiple linear regression.
Explore Association Between Pharmacokinetic Maximum Dose Concentration and disease Appropriate Circulating Tumor Marker PSA | Day 28
  The association between pharmacokinetic maximum dose concentration time and pharmacodynamic circulating tumor marker PSA will be assessed by multiple linear regression.
Explore Association Between Pharmacokinetic Maximum TCRT ESO A2 Dose Concentration Time and Pharmacodynamic Adverse Events as Identified by CTCAE Version 5. | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year.
  The association between pharmacokinetic parameters and pharmacodynamic adverse event incidence will be assessed by rank correlation.
Explore Association Between Pharmacokinetic Maximum Dose Concentration time and Pharmacodynamic Adverse Event Incidence. | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year.
  Explore association between pharmacokinetic maximum dose concentration time and pharmacodynamic adverse event incidence.
Explore Association Between Pharmacokinetic Maximum Dose Concentration and Area Under the Curve zero to infinity | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year.
  The association between maximum tolerated dose and area under the curve zero to infinity will be assessed by multiple linear regression.
Explore Pharmacokinetic Relationship with Tlast of CD3-positive/tetramer-positive T cells | Day -7, 1,2,3, 4, 5, 8,15, 28, 60, 90, 180, 270 and every 3 months until disease progression averaging one year.
  The association between pharmacokinetic parameters and [variable] will be assessed by multiple linear regression.
Explore Pharmacokinetic Relationship with Phenotype of Genetically Modified T cells in vivo | Baseline to disease progression averaging one year
  The association between pharmacokinetic parameters and phenotype of genetically modified T cells in vivo will be assessed by multiple linear regression.
Explore Pharmacokinetic Relationship with Tumor Objective Response Rate by RECIST 1.1 | 3 months
  The association between pharmacokinetic parameters and objective response rate will be assessed by multiple linear regression.
Explore Pharmacokinetic Relationship with Progression-Free Survival by RECIST 1.1 | 3 months
  The association between pharmacokinetic parameters and progression-free survival will be assessed by multiple linear regression.
Explore Pharmacokinetic Relationship With Disease Control Rate RECIST 1.1 | 3-months
  The association between pharmacokinetic parameters and disease control rate will be assessed by multiple linear regression
Explore Pharmacokinetic Relationship With Overall Survival RECIST 1.1 | Baseline to disease progression averaging one year
  The association between pharmacokinetic parameters and overall survival will be assessed by multiple linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Becerra, MD, Principal Investigator — Baylor University Medical Cancer Hospital

IPD SHARING:
Plan to Share IPD: No
No patients enrolled therefore no data available to share.